CLINICAL TRIAL: NCT03785223
Title: A 14 Week, Randomized, Placebo-Controlled Cross-Over Study of Methylphenidate Hydrochloride Controlled Release Capsules in Adult ADHD With and Without Anxiety Disorder Comorbidity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Purdue Pharma, Canada (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 5748
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Attention Deficit Hyperactivity Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Agoraphobia
Keywords: ADHD; Anxiety Disorders; Stimulants; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Agoraphobia; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylphenidate Hydrochloride Controlled-Release Capsules (Experimental): Flexibly dosed at 25-100 mg per day
  Interventions: Drug: Methylphenidate Hydrochloride Controlled-Release Capsules
- Placebo Capsules (Placebo Comparator): 1-4 capsules daily
  Interventions: Drug: Placebo Capsule

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride Controlled-Release Capsules — 25 mg methylphenidate hydrochloride- titrated as tolerated up to a maximum 4 capsules daily (25 mg- 100 mg total dose)
  At Week 0 or Week 7, dosing will start at 1 capsule/day for one week, and be titrated to 2 capsules/day for Week 2. 50 mg of methylphenidate hydrochloride per day (i.e. 2 capsules/day) is the minimum dose that must be achieved. The dose may be titrated to 75 mg/day for Week 3 and to 100 mg/day for Week 4 if participants are tolerating their current dose, are experiencing no adverse events, and have not fully responded. By Week 4 or Week 11, no further dose changes will occur.
  Other Names: Foquest
  Arms: Methylphenidate Hydrochloride Controlled-Release Capsules
Drug: Placebo Capsule — At Week 0 or Week 7, dosing will start at 1 capsule/day for one week, and be titrated to 2 capsules/day for Week 2. The dose may be titrated to 75 mg/day for Week 3 and to 100 mg/day for Week 4 if participants are tolerating their current dose, are experiencing no adverse events, and have not fully responded. By Week 4 or Week 11 no further dose changes will occur.
  Arms: Placebo Capsules

SUMMARY:
Other psychiatric disorders, including anxiety, often co-occur with adult ADHD; with 85% of ADHD patients having at least one other psychiatric condition. The presence of a co-occurring anxiety disorder has been associated with additive clinical effects, leading to more global impairment, poorer outcome, greater resistance to treatment and increased costs of illness. Stimulants are effective first-line treatments for adult ADHD patients, however the literature has mostly examined these treatments in pure ADHD populations (i.e. without other psychiatric disorders). Thus, there is little information to guide physicians in making treatment decisions for patients with ADHD and a co-occurring condition.

This trial aims to evaluate the efficacy and safety of methylphenidate hydrochloride controlled release capsules (Foquest) in treating adults aged 18-65 years with DSM-5 ADHD with and without a co-occurring anxiety disorder.The study uses a 14-week, randomized, placebo-controlled, cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient men and women between 18 and 65 years who meet criteria for Current DSM-5 ADHDalone or with one of the following DSM-5 diagnoses: GAD, SAD,PD or Agoraphobia. Major Depressive Disorder or Persistent Depressive Disorder will be allowed, providing the severity is considered moderate or less, as defined by a score on the Montgomery Depressive Rating Scale-MADRS score of ≤ 25.
2. ADHD rating scale for DSM-5 (ADHD-5-RS) score ≥ 24.
3. Concomitant treatment with selective serotonin reuptake inhibitors (SSRI's), serotonin noradrenaline reuptake inhibitors (SNRI's), benzodiazepines, beta-blockers, atypical anti-psychotics, anti-epileptics is allowed, provided the dose has been stable for 8 weeks prior to study entry. Dose changes of allowed concomitant medication should be avoided during the treatment phases of the study.
4. The ability to comprehend and satisfactorily comply with protocol requirements.
5. Written informed consent given prior to entering the baseline period of the study.
6. All women of child bearing potential must have a negative screening visit serum or urine pregnancy test and be using adequate contraception for the duration of the study. Medically acceptable forms of contraception include oral contraceptives, injectable or implantable methods, intrauterine devices or properly used barrier contraception. Additionally, the use of condoms is suggested as an adjunct to the methods previously addressed to provide additional protection against accidental pregnancy.

Exclusion Criteria:

1. Participants who currently fulfill criteria for a lifetime history of bipolar disorder, schizophrenia or other psychotic disorders, delirium, dementia and amnesic and other cognitive disorders, severe head injury, autism spectrum disorders, or are in a current agitated state.
2. Participants with a history of seizure disorders, or an unstable medical condition will also be excluded.
3. Participants with significant suicidal ideation (MADRS item 10 score > 3) or who have enacted suicidal behaviours within 6 months prior to intake will be excluded from study participation and referred for appropriate clinical intervention.
4. Current treatment with a stimulant.
5. A history of > 2 failed trials of adequately dosed psychostimulants for Adult ADHD.
6. Patients receiving current psychotherapy, including cognitive behavioural therapy for either ADHD or an anxiety disorder, within 4 weeks prior to the baseline period.
7. Patients who are known to be allergic to methylphenidate or components of methylphenidate hydrochloride, have known hypersensitivity or idiosyncrasy to methylphenidate hydrochloride.
8. Patients who have thyroid pathology, treatment of which has not been stabilized for at least 3 months.
9. MAO inhibitors within 3 weeks of the start of the baseline.
10. Individuals meeting criteria for current cannabis use disorder or substance use disorder will be excluded.
11. Current use of bupropion or tri-cyclic antidepressants, with the exception of clomipramine.
12. Current use of clonidine, modafinil or atomoxetine.
13. Previous intolerance or failure to respond to an adequate trial of methylphenidate hydrochloride controlled release capsules (defined as a minimum of 55mg per day for at least 4 weeks).
14. Patients who have a history or evidence of a medical condition that would expose them to an increase or significant adverse event or interfere with assessments of safety and efficacy during the course of the trial including: advanced arteriosclerosis, symptomatic cardiovascular disease, moderate to severe hypertension, or other pre-existing cardiac abnormalities or other serious cardiac problems.
15. Patients with a history of Glaucoma.
16. Sleep medications during the study period are excluded with the exception of zopiclone and zolpidem and melatonin.
17. Patients using any herbal psychoactive treatments, eg; St.John's Wort, Valerian, Kava Kava, or Chamomile Extract within 14 days prior to randomization.
18. Patients who have received electroconvulsive therapy within the previous 6 months.
19. Patients with any condition or on any therapy that in the investigator's opinion or as indicated in the methylphenidate hydrochlorideproduct label, that may pose a risk to the subject or interfere with the study objective.
20. Patients having clinically significant abnormal laboratory or ECG findings not resolved by the baseline examination.
21. Patients with a proximal family history of sudden, unexplained cardiac death.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-04-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Attention Deficit and Hyperactivity Rating Scale - 5 | Change from baseline to Week 12
  The ADHD-RS-5 is a scale for children and adolescents that assesses the frequency and severity of ADHD symptoms and impairments based on criteria from the Diagnostic Statistics Manual 5. The measure will be adapted for use with adults as a clinician rated scale in this study. It consists of 18 items, rated on a 4-point scale from 0 (never or rarely) to 3 (very often). The items can be summed to obtain a total score (range: 0-54), an Inattention subscore (range:0-27), and a Hyperactivity-Impulsivity subscore (range: 0-27), with higher scores indicating greater frequency and severity of symptoms.

SECONDARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | Change from baseline to Week 12
  The 14-item HAM-A was developed to assess general anxiety symptoms in a clinical population and has proven sensitive to change with treatment. It is a clinician-rated measure and will be administered by a trained, blinded rater, using the Structured Interview Guide for the HAM-A. It has 14-items to rate the intensity of psychic and somatic anxiety on a 5-point severity scale. Each item ranging from 0 (not present) to 4 (very severe) are summed up to give a total possible score of 0 (not present) to 56 (very severe), where lower scores indicates less anxiety.
Clinical Global Impression - Severity (CGI-S) | Change from baseline to Week 12
  The CGI-S is a clinician-rated instrument used to assess global severity of symptoms. The CGI-S ranges from 1 (normal, not ill) to 7 (among the most severely ill).
Clinical Global Impression - Improvement (CGI-I) | Change from baseline to Week 12
  The CGI-I is a clinician-rated instrument used to assess overall improvement of illness. The CGI-I ranges from 1 (very much improved) to 7 (very much worse).
Montgomery-Åsberg Depression Rating Scale (MADRS) | Change from baseline to Week 12
  The MADRS is a clinician rated scale evaluating depressive symptoms. It consists of 10 items assessed on a 7-point scale (range: 0-6). The total score ranges from 0 to 60, with higher scores indicating greater severity of depressive symptoms.
Barkley Adult ADHD Rating Scale (BAARS-IV) | Change from baseline to Week 12
  Self-report scale evaluating ADHD symptoms. Symptom count scores range from 1 to 27, with higher scores indicating more ADHD symptoms. Total scores range from 27 to 108, with higher scores indicating greater severity of symptoms.
Weiss Functional Impairment Rating Scale-Self Report (WFIRS-S) | Change from baseline to Week 12
  The WFRIS is a self-reported measure of functional impairment associated with ADHD in various clinically-relevant domains of functioning. It examines both symptoms and behviours or emotional problems that may have impacted each functioning in each domain. It consists of 70 items, rated on a 4-point scale from 0 (never or not at all) to 3 (very often or very much). Total scores range from 0 to 210, with higher scores indicative of greater ADHD-related functional impairment. Subscores may be calculated for specific domains by summing the items within that section: family (range: 0-24), work (range: 0-33), school (range: 0-33), life skills (range: 0-36), self-concept (range: 0-15), social (range: 0-27), and risk (range: 0-42).
Barkley Deficits in Executive Functioning Scale (BDEFS) | Change from baseline to Week 12
  The BDEFS is an adult self-report measure of executive functioning skills in daily life activities. It contains 20 items assessed on a 4-point scale ranging from 1 (never or rarely) to 4 (very often). The total score ranges from 20-80, with higher scores indicating greater deficit in executive functioning skills relevant to daily activities.
Overall Anxiety Severity and Impairment Scale (OASIS) | Change from baseline to Week 12
  The OASIS is a self-report measure assessing the severity and impairment associated with anxiety disorders. It contains 5 items rated on a 5-point scale (range: 0-4). The total score ranges from 0-20, with greater scores indicating greater severity of anxiety and related impairment.
Obsessive Compulsive Inventory - Revised (OCI-R) | Change from baseline to Week 12
  The OCI-R is a self-report scale for assessing symptoms of Obsessive-Compulsive Disorder (OCD). It consists of 18 questions with a 5-point scale (range: 0 to 4). The possible range of scores is 0 to 72, with higher scores indicating a greater likelihood of the presence of OCD.
Quick Inventory of Depressive Symptoms (QID-SR-16) | Change from baseline to Week 12
  The QIDS is a self-report measure of depression. It contains 16 items with a 4-point scale (range: 0 to 3) which assess the severity of the nine diagnostic symptom criteria used in the DSM: Sleep disturbance, sad mood, decrease/increase in appetite/weight, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, and psychomotor agitation/retardation. The total possible score is ranged from 0 to 27, with higher scores representing greater severity of depression.
Sheehan Disability Scale (SDS) | Change from baseline to Week 12
  The SDS is a 3 question instrument designed to assess functional impairment associated with mental disorders in three domains: work impairment, social impairment, and impairment of family life or home responsibilities. Each sub-scale score ranges from 0 to 10 and a total disability score, calculated as the sum of scores for each question ranges from 0 to 30. Higher scores reflect greater impairment.
Social Phobia Inventory (SPIN) | Change from baseline to Week 12
  The SPIN is a self-report questionnaire measuring the severity of social anxiety symptoms. It consists of 17 items assessed on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). The total possible score ranges from 0-68, with higher scores representing greater severity of social anxiety symptoms.
Generalized Anxiety Disorder-7 | Change from baseline to Week 12
  The GAD-7 is a self-reported questionnaire that measures the severity of various signs of GAD. It contains seven items with a 4-point scale (range: 0 to 3). The total possible score is ranged from 0 to 21, with higher scores representing greater severity of GAD.
Panic and Agoraphobia Scale (PAS) | Change from baseline to Week 12
  The PAS is a measure of the severity of illness in patients with panic disorder (with or without agoraphobia). It has 13 items with a 5-point scale (range: 0-4). The total possible score is ranged from 0 to 52, with higher scores representing increased severity of illness. It contains 5 sub-scales: panic attacks, agoraphobic avoidance, anticipatory anxiety, disability, and functional avoidance (health concerns).
PTSD Checklist for DSM-5 (PCL-5) | Change from baseline to Week 12
  The PCL-5 is a 20 item self-report measure that assesses symptoms of PTSD. Each item is rated on a 5-point scale from 0 (not at all) to 4 (extremely). The possible range of scores is 0 to 80, with higher scores indicating greater severity of PTSD.
Drug Abuse Screening Test (DAST) | Change from baseline to Week 12
  The DAST is a self-report measure used to identify individuals that are abusing drugs (not including alcohol). It contains 20 items requiring a "yes" or "no" response, of which "yes" is scored as 1 and "no" is scored as 0 for 18 items, and "yes" is scored as 0 and "no" is scored as 1 for 2 items. The total score ranges from 0-20, with higher scores indicated a greater degree of drug use and misuse issues.
Alcohol Use Disorders Identification Test (AUDIT) | Change from baseline to Week 12
  The AUDIT is a self-report screening test that assesses alcohol consumption, drinking behaviours, and alcohol-related problems. It consists of 20 items, 8 of which are rated on a 4-point scale from 0-4, and 2 of which are rated on a 3-point scale from 0, 2 and 4. The items are summed to obtain a total score ranging from 0-40, with higher scores indicating a greater degree of risky drinking. Consumption and dependance subscores (range: 0-12) may also be calculated by summing specific items.
Cannabis Use Disorder Identification Test-Revised (CUDIT-R) | Change from baseline to Week 12
  The CUDIT-R is a self-report screening test that assesses cannabis use and related problems. It contains 8 items, 7 of which are rated on a 5-point scale ranging from 0 (never) to 4 (daily or almost daily), and 1 of which is rated on a 3-point scale from 0, 2 and 4. The total score ranges from 0-32, with higher scores indicating more hazardous cannabis use.
Hoarding Rating Scale (HRS) | Change from baseline to Week 12
  The HRS will be administered as a self-report questionnaire to assess hoarding symptoms. It consists of 5 items rated on a 9-point scale from 0 (none) to 8 (extreme). The total scores range from 0-40, with greater scores indicating greater hoarding severity.
Binge Eating Scale (BES) | Change from baseline to Week 12
  The BES is a self-report measure of behaviours, cognitions, and emotions related to binge eating. It consists of 16 items, 14 of which are rated on a 4-point scale from 0-3, and 2 of which are rated on a 3-point scale from 0-2. The total score ranges from 0-46, with higher scores indicating more severe binge eating problems.
Pittsburgh Sleep Quality Index (PSQI) | Change from baseline to Week 12
  The PSQI is a self-report questionnaire which measures sleep quality, patterns, and disturbances. It consists of 9 items, 4 of which are rated on a 4-point scale of 0 (not during the past month) to 3 (3 or more times a week), and 1 of which is rated on a 4 point scale of 0 (very good) to 3 (very bad). The other 4 questions collect information on sleep time and duration. The items are summed to produce 7 component scores ranging from 0-3, which are subjective sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. These component scores are then combined to get the total score ranging from 0-21, with higher scores indicating worse sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Van Ameringen, MD, FRCPC, Principal Investigator — McMaster University
Locations (1):
- MacAnxiety Research Center, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided